CLINICAL TRIAL: NCT03411538
Title: A Prospective Surveillance Study for Outcome and Risk Factors Associated With Antibiotic-resistant Infections Among Patients With Hospital-acquired Infections
Brief Title: Mortality Related to AMR in Patients With Hospital-acquired Infection
Acronym: HAMR
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Sanpasitthiprasong Hospital (Other Government); Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Other Study IDs: MICRO1707
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2018-07

CONDITIONS: Hospital-acquired Infections
Keywords: antibiotic-resistant infections; risk factors; prospective surveillance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospital-acquired bacterial infection
  Interventions: Other: Collect data on clinical history

INTERVENTIONS:
Other: Collect data on clinical history — Collect data on clinical history, clinical manifestation, comorbidity, admission data, use of invasive medical intervention, history of antibiotic treatment and antibiotic susceptibility test results

SUMMARY:
This is a prospective surveillance study to estimate excess deaths due to and risk factors associated with antibiotic-resistant infection among patients with hospital-acquired infection (HAI) in a resource-limited setting. We will focus on six pathogenic bacteria that are of clinically important in the hospital.

DETAILED DESCRIPTION:
We will first identify patients with pathogenic bacteria isolated from clinical sample collected >48 hours after admission. These patients will then be screened for eligibility criteria. Signed informed consent will be sought from the enrolled patients. The primary outcome is survival status within 28 days since the first specimen culture positive for one of the six organisms of interest. All patients with hospital-acquired infection will be assessed for in-hospital 28-day survival as part of the routine hospital surveillance system. Follow-up to confirm 28-day outcome via telephone call will be performed only if patient signed informed consent and permission is granted. All isolates from positive cultures will be collected and stored securely.

This study will not interfere with standard patient care or routine diagnosis procedure, hence subject will receive no direct medical harm or benefits from being in the study. Researchers of this study will not be involved in the management, care and treatment of study subjects. Patient care will remain under the responsibility of the attending medical staff according to standard practice of care. The study team will work closely with the hospital Infectious Control team to screen and enroll patients as part of the HAI surveillance data system in Sunpasitthiprasong Hospital. This study will be an enhancement of the current HAI surveillance system, which will provide data on 28-day survival status, Charlson Comorbidities Index (CCI) score and Sequential Organ Failure Assessment (SOFA) score for each patient and risk factors related to acquiring hospital-acquired infection to the hospital Infectious Control (IC) team.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any age admit at Sunpasitthiprasong Hospital
* At least one of the six organisms, which include Staphylococcus aureus, Enterococcus spp., Escherichia coli, Klebsiella pneumoniae, Pseudomonas aeruginosa, Acinetobacter spp., isolated from clinical specimen >48 hours after admission
* Acquired Bloodstream infection (BSI), Lower-respiratory tract infection(LRTI), Skin/Soft tissue infection (SSTI), Surgical-site infection (SSI), Urinary tract infection (UTI) or infection at other body sites >48 hours after admit at the hospital

Exclusion Criteria:

• Clinical symptoms of current infection presented ≤48 hours of admission

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target study subjects include male and female patients of any age admit at the hospital, and acquired hospital-acquired bacterial infection during hospital stay. We will focus on six key pathogens that were in the WHO global priority list of antibiotic-resistant bacteria and are also of clinical importance in resource-limited settings, namely:
  * Staphylococcus aureus
  * Enterococcus spp
  * Escherichia coli
  * Klebsiella pneumoniae
  * Pseudomonas aeruginosa
  * Acinetobacter spp
  The severity of underlying illness will be assessed using Charlson Comorbidity Index (CCI) score and severity of the infection will be assessed using Sequential Organ Failure Assessment (SOFA) score. These score will be reported to the physician whenever appropriate.
Sampling Method: Probability Sample
Enrollment: 2069 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Assoc. Prof. Direk Limmathurotsakul, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Sunpasitthiprasong Hospital, Ubon Ratchathani, Thailand

REFERENCES:
- [Derived] Lim C, Teparrukkul P, Nuntalohit S, Boonsong S, Nilsakul J, Srisamang P, Sartorius B, White NJ, Day NPJ, Cooper BS, Limmathurotsakul D. Excess Mortality Attributable to Hospital-Acquired Antimicrobial-Resistant Infections: A 2-Year Prospective Surveillance Study in Northeast Thailand. Open Forum Infect Dis. 2022 Jun 20;9(9):ofac305. doi: 10.1093/ofid/ofac305. eCollection 2022 Sep. PMID 36092827